CLINICAL TRIAL: NCT04208048
Title: Post-market Surveillance Study of FLXfitTM 15 TLIF Interbody Fusion Device
Brief Title: FLXfitTM 15 TLIF Interbody Fusion Device
Status: Completed | Type: Observational
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Kern Singh, MD, Attending Orthopedic Surgeon, Rush University Medical Center
Other Study IDs: 18073011
Record Dates: First submitted 2019-09-06; First posted 2019-12-23 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Degenerative Disc Disease
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- FLXfit 15: The FLXfit 15 device will then be placed into the space between the low backbones, using specific medical instruments, where the damaged disc was removed.
  Interventions: Device: FLXfit 15TM device

INTERVENTIONS:
Device: FLXfit 15TM device — In order to implant the FLXfit 15TM device properly, your study doctor will first prepare the space between the low back bones (vertebrae) and then remove your damaged disc. The FLXfit 15TM device will then be placed into the space between the low backbones, using specific medical instruments, where the damaged disc was removed.

SUMMARY:
The purpose of this study is post-market, patient outcome research to evaluate medical device safety and effectiveness. The data collected will assess the safety of the FLXfit 15TM (studydevice) system.

DETAILED DESCRIPTION:
The purpose of this study is post-market, patient outcome research to evaluate medical device safety and effectiveness. The data collected will assess the safety of the FLXfit 15TM (study device) system, as measured by the rate of serious operative and post-operative complications. It will also assess the effectiveness as measured by radiographs (X-rays), CT scans, MRI scans, patient-reported, health-related quality of life questionnaires up to (24) months following the procedure, as compared to before surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18-70 y/o)
* Male or Female
* With the following conditions of the lumbar spine as confirmed by advanced imaging (CT or MRI), who is a candidate for primary spinal fusion procedure according to acceptable criteria for such medical conditions:

  * Degenerative disc disease with up to Grade I spondylolisthesis
  * Spondylolisthesis
* Failure of at least 6-months conservative treatment
* BMI < 40
* Patient to approve no pregnancy during the 24 months of study and no participation in other studies in parallel to this one
* Ability to read, understand, and sign informed consent

Exclusion Criteria:

* Infection, local to the operative site
* Signs of local inflammation
* Fever or leukocytosis
* Pregnancy
* Significant mental disorder or condition that could compromise the patient's ability to remember and comply with preoperative and postoperative instructions (e.g. current treatment for a psychiatric/psychosocial disorder, senile dementia, Alzheimer's disease, traumatic head injury)
* Prior surgical procedure (with the exception of decompression only procedure) at the index level(s) using the desired operative approach
* Prior fusion procedure at an adjacent level
* Any other condition which would preclude the potential benefit of spinal implant surgery, such as the presence of tumors or congenital abnormalities, fracture local to the operating site, elevation of segmentation rate unexplained by other diseases, elevation of white blood count (WBC), or a marked left shift in the WBC differential count
* Neuromuscular disorder that would engender unacceptable risk of instability, implant fixation failure, or complications in postoperative care
* Active local infection in or near the operative region
* Active systemic infection and/or disease
* Severe osteoporosis or insufficient bone density, which in the medical opinion of the physician precludes surgery or contraindicates instrumentation
* Endocrine or metabolic disorders known to affect osteogenesis (e.g. Paget's disease, renal osteodystrophy, hypothyroidism)
* Systemic disease that requires the chronic administration of nonsteroidal anti- inflammatory or steroidal drugs
* Suspected or documented allergy or intolerance to implant's materials
* Symptomatic cardiac disease
* Patient unwilling to cooperate with postoperative instructions.
* Any case where the implant components selected for use would be too large or too small to achieve a successful result.
* Patient having inadequate tissue coverage over the operative site or inadequate bone stock or quality.
* Any patient in which implant utilization would interfere with anatomical structures or expected physiological performance.
* Prior fusion at the level to be treated.
* Back VAS < 4/10

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with degenerative disc disease (DDD) at one or two contiguous levels from L2 to S1. Patients may also have up to Grade I spondylolisthesis or retrolisthesis at the involved level(s). Patients should be skeletally mature and have completed six months of non-operative treatment.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-08-22 (Actual)

PRIMARY OUTCOMES:
Fusion | through study completion; 2 year
  Did patient achieve fusion?
Visual Analogue Pain Scale: Back | 6-week
  0 to 10 score; higher score means worse pain
Visual Analogue Pain Scale: Back | 12- week
  0 to 10 score; higher score means worse pain
Visual Analogue Pain Scale: Back | 6-month
  0 to 10 score; higher score means worse pain
Visual Analogue Pain Scale: Back | 1-year
  0 to 10 score; higher score means worse pain
Visual Analogue Pain Scale: Back | 2-year
  0 to 10 score; higher score means worse pain
Visual Analogue Pain Scale: Leg | 6-week
  0 to 10 score; higher score means worse pain
Visual Analogue Pain Scale: Leg | 12- week
  0 to 10 score; higher score means worse pain
Visual Analogue Pain Scale: Leg | 6-month
  0 to 10 score; higher score means worse pain
Visual Analogue Pain Scale: Leg | 1-year
  0 to 10 score; higher score means worse pain
Visual Analogue Pain Scale: Leg | 2-year
  0 to 10 score; higher score means worse pain
Oswestry Disability Index | 6-week
  0 to 100 score; higher score means greater patient disability
Oswestry Disability Index | 12- week
  0 to 100 score; higher score means greater patient disability
Oswestry Disability Index | 6-month
  0 to 100 score; higher score means greater patient disability
Oswestry Disability Index | 1-year
  0 to 100 score; higher score means greater patient disability
Oswestry Disability Index | 2-year
  0 to 100 score; higher score means greater patient disability
Short Form-12 Health Survey | 6-week
  0 to 100 score; higher score means less patient disability
Short Form-12 Health Survey | 12-week
  0 to 100 score; higher score means less patient disability
Short Form-12 Health Survey | 6-month
  0 to 100 score; higher score means less patient disability
Short Form-12 Health Survey | 1-year
  0 to 100 score; higher score means less patient disability
Short Form-12 Health Survey | 2-year
  0 to 100 score; higher score means less patient disability
Patient Reported Outcomes Measurement Information System (PROMIS) | 6-week
  20 to 80 score; higher score means higher reported self-capability
Patient Reported Outcomes Measurement Information System (PROMIS) | 12- week
  20 to 80 score; higher score means higher reported self-capability
Patient Reported Outcomes Measurement Information System (PROMIS) | 6-month
  20 to 80 score; higher score means higher reported self-capability
Patient Reported Outcomes Measurement Information System (PROMIS) | 1-year
  20 to 80 score; higher score means higher reported self-capability
Patient Reported Outcomes Measurement Information System (PROMIS) | 2-year
  20 to 80 score; higher score means higher reported self-capability

CONTACTS AND LOCATIONS:
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
All study related documents will be shared through a password protected and encrypted program managed by Midwest Orthopedics IT department.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will become available after the participant has signed the informed consent and will remain available until the study is closed.
Access Criteria: The study staff will have to complete HIPPA and confidentiality training. In addition, they must by Midwest Orthopedics staff who will access the information on a password protected and encrypted computer.

DOCUMENTS (1):
  • Informed Consent Form (2020-09-21): https://cdn.clinicaltrials.gov/large-docs/48/NCT04208048/ICF_001.pdf